CLINICAL TRIAL: NCT05626543
Title: The Effect of Mindfulness-based Cognitive Behavior Therapy on Occupational Stress Management Among Community Secondary School Teachers in Kathmandu
Brief Title: The Effect of Mindfulness-based Cognitive Behavior Therapy on Occupational Stress Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University (Other)
Responsible Party: Principal Investigator, Subas Neupane, Study director, Tampere University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 147
Record Dates: First submitted 2022-11-09; First posted 2022-11-23 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Occupational Stress
Keywords: Occupational stress; Schoolteachers; mindfullness; Cognitive behavior
MeSH Terms: conditions — Occupational Stress | interventions — Cognitive Behavioral Therapy; Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: Cognitive behavior therapy (CBT) and Mindfulness-based stress reduction (MBSR) programs will be used together.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in the Intervention arm will receive Cognitive behavior therapy (CBT) and Mindfulness-based stress reduction (MBSR) programs based intervention.
  Interventions: Behavioral: Cognitive behavior therapy (CBT) and Mindfulness-based stress reduction (MBSR) programs
- Control (No Intervention): The control will work normally with intervention. The intervention material will be provided to the controls once the follow-up surveys are conducted after the intervention is given to the intervention arm.

INTERVENTIONS:
Behavioral: Cognitive behavior therapy (CBT) and Mindfulness-based stress reduction (MBSR) programs — Cognitive behavior therapy (CBT) and Mindfulness-based stress reduction (MBSR) programs will be used combinedly. CBT will be constructed based on the CBT model of Beck, (2021) and mindfulness practice will be implemented based on the MBSR program developed by Williams et. al. (2011).
  Arms: Intervention

SUMMARY:
Occupational stress is one of the leading work-related factors that influence the health of employees and their ability to work. Stress at work is unavoidable due to changing and increasing demands and types of work. The teaching profession is one of the most stressful jobs with a high level of psychological morbidity globally. Stress may occur together with common mental disorders, which are one of the leading causes of disability worldwide. However, very little is known about the occurrence of occupational stress among schoolteachers. Several interventions have been designed to help school teachers to cope with stress. However, lifestyle modification intervention is not well explored, therefore, this study aims to evaluate the impact of lifestyle modification intervention on occupational stress management among community-level schoolteachers. Through effective intervention tools, workplace health can be enhanced, and the well-being of schoolteachers could be maintained.

DETAILED DESCRIPTION:
Background

Stress is the feeling of being overwhelmed or unable to cope with mental or emotional pressure which can happen together with mental health problems, such as depression. In 2019, depressive disorders were the sixth leading contributor to disability-adjusted life years (DALYs) among 25-49-year-olds. Occupational stress is the most common form of stress, and the degree of stress varies among different occupations. A study from the UK found that teaching was one of the most stressful occupations, because of its direct human-oriented nature. Likewise, a follow-up study in West England reported a higher level of psychological distress among a cohort of teachers than among comparable professionals from the general population.

Potential stressors for teachers are low job support, student apathy, overcrowded and noisy working environments, excessive paperwork, low wages, unsupportive parents, and changing curricula. Lacking management of chronic workplace stress may result in Burnout syndrome. Prolonged stress becomes permanent, over time, because it is hard to recover and as a result, the individual faces chronic fatigue, dementia, musculoskeletal problems, cardiovascular disease, and professional burnout syndrome. The range of job stress may vary from job to job and profession to profession. Largo-Wight, Moore, and Barr have shown some different roots of job stress pertaining to physical or biological and psychological or behavioral in nature. Notwithstanding, exploring the level of job stress in the working population, and their lifestyle modification practices to reduce the stress level have a significant implication. The large number of schoolteachers teaching at different levels may have multifaceted stresses due to various reasons, such as less pay, high job demands, job insecurity, lack of professional opportunity, and safety. An earlier study by Kumar et. al. stated that occupational stress is increasingly common in the teaching profession due to increased occupational complexities and economic pressure on individuals. The reason behind the increased distress among the teachers is the result of the failure of the school to meet the social needs and job demands of the teachers.

With most adults spending around half of their waking hours at work, the workplace is therefore an important setting to promote health and well-being. Various national and international bodies (e.g. ILO, WHO) are responsible for ensuring the health and safety of employees, with a focus on identifying physical, chemical, and biological hazards in the workplace. Increasingly, attention is also being paid to the psychosocial work environment, with a major focus on work stress. Therefore, promoting awareness of the link between stress and health among both employers and workers is an important component of workplace health promotion. Several interventions are tested to help teachers to reduce their stress levels and to improve their well-being and student outcomes at organizational and individual levels. Organizational-level interventions are directed at changing the organization's culture and work practices, whereas individual-level interventions are the most common approaches that include psychological relaxation or meditation, cognitive behavioral techniques to improve active coping skills, and lifestyle modification activities. Evidence shows that individual-level intervention improves teachers' health and well-being. In this regard, a study carried out by Naghieh et al. concluded that organizational interventions led to improvements in teacher well-being and retention rates. However, these lifestyle modification knowledge and practices have not been well explored among community-level schoolteachers. Therefore, this study aims to evaluate the impact of lifestyle modification intervention on occupational stress management among community-level schoolteachers. This individual-level intervention may affect teachers' own health behaviors, inspire others to review their own lifestyle activities, and support in developing a positive impact on community health practices.

Research aims and objectives

The overarching aim of this project is to investigate the effect of mindfulness-based cognitive behavior therapy on occupational stress management among secondary school teachers in Kathmandu, Nepal. The study has the following specific objectives:

* To assess the prevalence of occupational stress and the associated factors among schoolteachers.
* To evaluate the effect of the intervention on the occupational stress of teachers at post-intervention.
* To evaluate the effect of the intervention on the occupational stress of teachers in three months of follow-up after the intervention.

Subjects and methods

Study population and design: This research project plans to utilize an experimental study design focusing on community school settings and the prevailing numbers of teachers. Secondary-level teachers teaching at community schools from the Kathmandu district are the study population. The list of all schools in Kathmandu district (n=167) will be prepared and using 40 schools will be selected and 5 teachers from each school, totaling 200 teachers from these schools. Among them, teachers from 20 schools will be selected for the control group and another 20 will be for the intervention.

Sample size and power calculation: The estimated sample size will be proportional to the prevalence of occupational stress among schoolteachers. This study will try to use the power of 80%. There is a need for a sample of 90 teachers in each study group and 180 in total and assuming 10% attrition rate, the participants per study group will be 100 and in total 200 teachers.

Intervention: The content of the intervention has developed based on the previous literature. Cognitive behavior therapy (CBT) and Mindfulness-based stress reduction (MBSR) programs will be used combinedly.

Data collection tools:

The Maslach Burnout Inventory-Educators Survey (MBI-ES) will be used to measure the stress level of the teacher, as well as the effectiveness of intervention simultaneously. Demographic information of the participants will be collected using a separate set of questionnaires. The MBI-ES consists of 22 items including three sub-scales viz. Emotional Exhaustion (EE-9 items), Depersonalization (DP-5 items), and Personal Accomplishment (PA-8 items). These 22 items have different and unique values. The EE-9, and the DP-5, subscales, exhibit that the greater value the higher the stress they imply, however the PA-8 displays that the greater score the lower stress it indicates. The data collection will be carried out in three stages - at the baseline survey (T1), immediately after treatment (T2), and a follow-up measurement (T3) is scheduled for three months after the T2. The PI of the current project has prepared the first draft of the translation of this tool into the Nepali language. Two professional experts checked and corrected the translation of the tool. Further modifications in the tools will be carried out after using the tools for the pilot study and a final version will be prepared and ready for use.

Ethical considerations:

The permission to conduct this workplace intervention study has been taken from the concerned authorities and the ethical clearance was obtained from the Nepal Health Research Council (NHRC) (ethical approval number 147). Written/verbal consent was obtained from the study participants and their schools. In addition, the privacy and confidentiality of the participants will be maintained in the study according to scientific norms.

ELIGIBILITY:
Inclusion Criteria:

* In community schools, teachers who are employed at least one year before the survey and have a work contract of more than one year until the time of the survey;
* Teachers teaching in grades 9 and 10;
* Teacher of working age between 18 and 60 years;
* Teacher with any educational background and level; and
* Teacher who teaches any subjects at the secondary level (grades 9 and 10).

Exclusion Criteria:

* Teacher with a short-term contract (less than 1 year);
* Teacher employed for extra class or substitute;
* Currently pregnant or those are on maternity leave; and
* Teacher who is on study leave or absence due to long-term sickness.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 218 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Occupational stress | Baseline, change in the outcome will be assessed at post intervention (at 1 month), and in a 2 month of follow-up after the intervention
  Maslach Burnout Inventory-Educators Survey (MBI-ES) will be used to measure the outcome

CONTACTS AND LOCATIONS:
Overall Officials: Subas Neupane, Study Director — Tampere University; Netra Raj Paudel, Principal Investigator — Tampere University
Locations (1):
- Tampere University, Tampere, Pirkanmaa, Finland

IPD SHARING:
Plan to Share IPD: No
The data will be made available for others to use on request

REFERENCES:
- [Result] Ahola K, Salminen S, Toppinen-Tanner S, Koskinen A, Vaananen A. Occupational burnout and severe injuries: an eight-year prospective cohort study among Finnish forest industry workers. J Occup Health. 2013;55(6):450-7. doi: 10.1539/joh.13-0021-oa. Epub 2013 Oct 26. PMID 24162145
- [Result] Akanaeme IN, Ekwealor FN, Ifeluni CN, Onyishi CN, Obikwelu CL, Ohia NC, Obayi LN, Nwaoga CT, Okafor AE, Victor-Aigbodion V, Ejiofor TE, Afiaenyi IC, Ekomaru CI, Dike IC. Managing job stress among teachers of children with autism spectrum disorders: A randomized controlled trial of cognitive behavioral therapy with yoga. Medicine (Baltimore). 2021 Nov 19;100(46):e27312. doi: 10.1097/MD.0000000000027312. PMID 34797272
- [Result] GBD 2019 Diseases and Injuries Collaborators. Global burden of 369 diseases and injuries in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2020 Oct 17;396(10258):1204-1222. doi: 10.1016/S0140-6736(20)30925-9. PMID 33069326
- [Result] Wink G, Fransen G, Huisman M, Boersma S, van Disseldorp L, van der Velden K, Wagemakers A, van den Muijsenbergh M. 'Improving Health through Reducing Stress': Parents' Priorities in the Participatory Development of a Multilevel Family Health Programme in a Low-Income Neighbourhood in The Netherlands. Int J Environ Res Public Health. 2021 Jul 31;18(15):8145. doi: 10.3390/ijerph18158145. PMID 34360438
- [Result] Bernotaite L, Malinauskiene V. Workplace bullying and mental health among teachers in relation to psychosocial job characteristics and burnout. Int J Occup Med Environ Health. 2017 Jun 19;30(4):629-640. doi: 10.13075/ijomeh.1896.00943. Epub 2017 Apr 20. PMID 28584320
- [Result] Johnson S, Cooper C, Cartwright S, Donald I, Taylor P, Millet C. The experience of work-related stress across occupations. Journal of managerial psychology. 2005 Mar 1.
- [Result] Maslach, C., Leiter, M.P. (1999). Teacher burnout: A research agenda. In R. Vandenberghe & A. M. Huberman (Eds.), Understanding and preventing teacher burnout: A sourcebook of international research and practice. New York, NY: Cambridge University Press. 295-303.
- [Result] Titheradge D, Hayes R, Longdon B, Allen K, Price A, Hansford L, Nye E, Ukoumunne OC, Byford S, Norwich B, Fletcher M, Logan S, Ford T. Psychological distress among primary school teachers: a comparison with clinical and population samples. Public Health. 2019 Jan;166:53-56. doi: 10.1016/j.puhe.2018.09.022. Epub 2018 Nov 15. PMID 30448692
- [Result] Kumar, & Pragadeeswaran, S. (2011). Effects of occupational stress on spiritual quotient among executives. International Journal of Trade, Economics and Finance, Vol. 2 (4).
- [Result] Kivimaki M, Kawachi I. Work Stress as a Risk Factor for Cardiovascular Disease. Curr Cardiol Rep. 2015 Sep;17(9):630. doi: 10.1007/s11886-015-0630-8. PMID 26238744
- [Result] Gnawali, A. (2017). Work-Family balance and its outcome among female teachers in Nepal. International Journal of Research in Business Studies and Management Volume 4 (6), Pp. 23-29.
- [Result] Jennings, P. A., Brown, J. L., Frank, J. L., Doyle, S., Oh, Y., Davis, R., ... & Greenberg, M. T. (2017). Impacts of the CARE for Teachers program on teachers' social and emotional competence and classroom interactions. Journal of Educational Psychology, 109(7), 1010.
- [Result] Tsang KKY, Shum KK, Chan WWL, Li SX, Kwan HW, Su MR, Wong BPH, Lam SF. Effectiveness and Mechanisms of Mindfulness Training for School Teachers in Difficult Times: A Randomized Controlled Trial. Mindfulness (N Y). 2021;12(11):2820-2831. doi: 10.1007/s12671-021-01750-1. Epub 2021 Sep 16. PMID 34545293
- [Result] Greenberg, M.T., Brown, J.L., & Abenavoli, R. M. (2016). Teacher stress and health effects on teachers, students, and schools. Edna Bennett Pierce Prevention Research Center, Pennsylvania State University, 1-12.
- [Result] Naghieh A, Montgomery P, Bonell CP, Thompson M, Aber JL. Organisational interventions for improving wellbeing and reducing work-related stress in teachers. Cochrane Database Syst Rev. 2015 Apr 8;2015(4):CD010306. doi: 10.1002/14651858.CD010306.pub2. PMID 25851427
- [Derived] Paudel NR, Kc P, Ghimire R, Nygard CH, Neupane S. Occupational burnout and their determinants among schoolteachers in Nepal: a cross-sectional study. BMC Psychiatry. 2024 Jun 27;24(1):472. doi: 10.1186/s12888-024-05923-9. PMID 38937696
- See also: Mental Health Foundation, MHF. (2021). Stress. — https://www.mentalhealth.org.uk/a-to-z/s/stress